CLINICAL TRIAL: NCT03484832
Title: Comparison of the Effects of Vapocoolant Spray and Topical Anesthetic Cream on Pain During Intra-articular Injection of Shoulder
Brief Title: Spray vs EMLA Cream on Pain During Intra-articular Injection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, SANGHYUN KIM, MD. PhD. Professor of Physical Medicine and Rehabilitation, Soonchunhyang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMLA SPRAY
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Adhesive Capsulitis of the Shoulder
MeSH Terms: conditions — Bursitis | interventions — Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Spray group (Experimental): Using Walter Ritter Ethyl Chloride Spray and placebo cream
  Interventions: Device: Walter Ritter Ethyl Chloride Spray; Other: Placebo Cream
- EMLA group (Experimental): Using EMLA cream and placebo spray
  Interventions: Other: Placebo Spray; Drug: EMLA Cream
- Placebo group (Placebo Comparator): Using placebo cream and placebo spray
  Interventions: Other: Placebo Spray; Other: Placebo Cream

INTERVENTIONS:
Device: Walter Ritter Ethyl Chloride Spray — Participants receive an application of EMLA or placebo cream at the needle electrode insertion site 60 minutes before needle insertion, and a self adhering dressing is placed over the site. After 60 minutes, the dressing and cream are removed from the site, then the insertion site is sprayed from a distance of 30 cm for 5 seconds or until the skin was blanched, then intra-articular injection of shoulder is performed.
  Arms: Spray group
Other: Placebo Spray — Participants receive an application of EMLA or placebo cream at the needle electrode insertion site 60 minutes before needle insertion, and a self adhering dressing is placed over the site. After 60 minutes, the dressing and cream are removed from the site, then the insertion site is sprayed using placebo spray (Evain Eau Minerale Naturelle, a pure water spray with hydrocarbon propellant), then intra-articular injection of shoulder is performed.
  Arms: EMLA group; Placebo group
Other: Placebo Cream — Participants receive an application of placebo cream at the needle electrode insertion site 60 minutes before needle insertion, and a self adhering dressing is placed over the site. After 60 minutes, the dressing and cream are removed from the site, then the insertion site is sprayed using Walter Ritter Ethyl chloride spray or placebo spray, then intra-articular injection of shoulder is performed.
  Arms: Placebo group; Spray group
Drug: EMLA Cream — Participants receive an application of EMLA cream at the needle electrode insertion site 60 minutes before needle insertion, and a self adhering dressing is placed over the site. After 60 minutes, the dressing and cream are removed from the site, then the insertion site is sprayed using Walter Ritter Ethyl chloride spray or placebo spray, then intra-articular injection of shoulder is performed.
  Other Names: EMLA 5% cream
  Arms: EMLA group

SUMMARY:
All participants are randomly allocated to the spray group, EMLA group and placebo group. In spray group, participants receive an application of placebo cream at the needle electrode insertion site 60 minutes before needle insertion, and a self adhering dressing is placed over the site. After 60 minutes, the dressing and cream are removed from the site, then the insertion site is sprayed from a distance of 30 cm for 5 seconds or until the skin was blanched, then intra-articular injection of shoulder is performed. Immediately after injection, participants are asked to fill out the visual analog scale for injectional pain, five point Likert scale for satisfaction about the topical anesthesia. In EMLA group, participants receive an EMLA cream and placebo spray. In placebo group, participants receive a placebo cream and placebo spray.

DETAILED DESCRIPTION:
All participants are randomly allocated to the spray group, EMLA group and placebo group.

In spray group, participants receive an application of placebo cream at the needle electrode insertion site 60 minutes before needle insertion, and a self adhering dressing is placed over the site. After 60 minutes, the dressing and cream are removed from the site, then the insertion site is sprayed using ethyl chloride spray (Walter Ritter GmbH and Co., Hamburg, Germany) from a distance of 30 cm for 5 seconds or until the skin was blanched, then intra-articular injection of shoulder is performed. Immediately after injection, participants are asked to fill out the visual analog scale for injectional pain, five point Likert scale for satisfaction about the topical anesthesia.

In EMLA group, participants receive an application of EMLA cream at the needle electrode insertion site 60 minutes before needle insertion, and a self adhering dressing is placed over the site. After 60 minutes, the dressing and cream are removed from the site, then the insertion site is sprayed using placebo spray (Evain Eau Minerale Naturelle, a pure water spray with hydrocarbon propellant), then intra-articular injection of shoulder is performed. Immediately after injection, participants are asked to fill out the same scales.

In placebo group, participants receive a placebo cream and placebo spray.

ELIGIBILITY:
Inclusion Criteria:

* Who had a normative schedule of intra-articular injection of shoulder

Exclusion Criteria:

* those who refused to participate, those who were unable to understand a visual analog scale or a Likert scale, those with a history of an allergic reaction to vapocoolant spray or lidocaine, those with a history of cold intolerance (eg, Raynaud syndrome), those who took pain medications or had used topical anesthetics within the previous 24 hours, those with prior history of intra-articular injection of shoulder, those who exhibited an abnormal shoulder sensation on neurologic examination

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2018-03-14 (Actual); Primary Completion 2020-03-19 (Estimated); Study Completion 2020-05-19 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale for injection pain | Within 5 minute
  The 100-mm VAS consisted of a 100-mm horizontal line labeled ''no pain'' at the left and ''worst pain imaginable'' at the right.

SECONDARY OUTCOMES:
Five point Likert scale for participant's satisfaction | Within 5 minute
  The five-point Likert scale (1, strongly agree; 2, agree; 3, undecided; 4, disagree; and 5, strongly disagree) is used to answer the question: ''Are you satisfied with the topical anesthetic methods used before performing the shoulder intra-articular injection?''
Five point Likert scale for preferences for future usage | Within 5 minute
  The five-point Likert scale (1, strongly agree; 2, agree; 3, undecided; 4, disagree; and 5, strongly disagree) is used to answer the question: "Would you use the topical anesthetic methods applied today again if the shoulder intra-articular injection is repeated in the future?"

CONTACTS AND LOCATIONS:
Overall Officials: SANGHYUN KIM, Principal Investigator — Soonchunhyang University Hospital
Locations (1):
- Soonchunhyang University Hospital, Bucheon, Bucheon-si, Gyeonggido, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moon YE, Kim SH, Seok H, Lee SY. Comparison of the Effects of Vapocoolant Spray and Topical Anesthetic Cream on Pain During Intraarticular Injection of the Shoulder: A Randomized Double-Blind Controlled Trial. Arch Phys Med Rehabil. 2020 Oct;101(10):1689-1695. doi: 10.1016/j.apmr.2020.04.021. Epub 2020 May 20. PMID 32445850